CLINICAL TRIAL: NCT02247024
Title: Dynamic Assessment of Pupillary Reflex in Patients on High-dose Opioids
Brief Title: Pupil Response in Patients on Opioids.
Acronym: Pupillometry
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ulf Kongsgaard, Professor, Oslo University Hospital
Other Study IDs: 2014/1226
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2018-10

CONDITIONS: Chronic Pain; Impaired Pupillary Reflex; Opioid-Related Disorders
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of pupillary reflex in patients on high-dose opioids. Clinical assessment of pain intensity, sedation score, and other side effects of opioids. Measurements of the concentration of opioids and their active metabolites in blood.

DETAILED DESCRIPTION:
Pupil size reflects the balance between sympathetic and parasympathetic systems. Pupil size and reaction are also influenced by drugs, where opioids result in miosis, an effect that is not considered to be influenced by opioid tolerance. However, cancer patients on high-dose opioids do not always present small pupil size.

We want to perform a dynamic assessment of pupillary reflex in patients on high-dose opioids. In addition to pupil size measurements under standard room light conditions, two pupil size reflexes will by assessed: the pupillary light reflex when the pupil is exposed to light, and the reflex dilation during a standardized noxious stimulus. On the same time we will assess pain intensity, sedation score, and other side effects of opioids while measuring the concentration of opioids and their active metabolites in blood. In addition we will register all concomitant medication that also might influence pupil size and reaction. Patients on more than 60 morphine equivalents pr day will be included.

ELIGIBILITY:
Inclusion Criteria:

* In-patients and out-patients at Oslo University Hospital with cancer pain who have use opioids (morphine, oxycodone, fentanyl or methadone or a combination of these drugs) at least for periods of 4 weeks, and use opioids corresponding to at least 60 mg oral morphine equivalents pr day

Exclusion Criteria:

* Patients who have undergone eye-surgery that may influence pupillary reflexes
* Patients on local medication that may influence pupillary reflexes
* Patients with amyloidosis, multiple sclerosis, Horner's syndrome, or ongoing migraine attack
* Patients with brain tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer pain on high-dose opioids; i.e. more than 60 morphine equivalents pr day
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2015-01; Primary Completion 2018-08 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Pupillary reflexes | One year
  Dynamic pupillometry

SECONDARY OUTCOMES:
Opioid and metabolite concentration | One year

CONTACTS AND LOCATIONS:
Overall Officials: Ulf E Kongsgaard, MD PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Oslo University Hospital, The Norwegian Radium Hospital, Oslo
  - The Norwegian Radium Hospital, Oslo

REFERENCES:
- [Derived] Kongsgaard UE, Hoiseth G. Dynamic assessment of the pupillary reflex in patients on high-dose opioids. Scand J Pain. 2019 Jul 26;19(3):465-471. doi: 10.1515/sjpain-2019-0032. PMID 31031265